CLINICAL TRIAL: NCT04343352
Title: Randomized Controlled Study: Evaluation of the Efficiency of Mobile Application for Parents of Children With Epilepsy
Brief Title: Evaluation of the Efficiency of Mobile Application for Parents of Children With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DILEK SAYIK (Other)
Responsible Party: Sponsor-Investigator, DILEK SAYIK, Principal Investigator, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSAYIK; Ayfer ACIKGOZ (Other: Eskisehir Osmangazı University); Sevgi YİMENİCİOĞLU (Other: Eskısehir City Hospıtal)
Record Dates: First submitted 2020-04-04; First posted 2020-04-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Child; Epilepsy; Education; Mobile Application; Nursing
Keywords: Child; Epilepsy; Parental Education; Mobile Application; Pediatric Nurse
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental study. Pretest - posttest with control and application group
Masking Description: Researchers and family will know about all the details of the study. Verbal and written permission will be obtained from families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In application group; Mobile Epilepsy Training Program Impleme (Experimental): * Mobile epilepsy training program will be introduced to the parents in the application group and pre-tests (Parent Epilepsy Knowledge Scale for Parents and Parental Anxiety Scale for Seizures Scale).
  * The participants will only use the mobile epilepsy training program application.
  * Parents in the application group will be monitored for 3 months using the mobile epilepsy training program. The researcher will follow the participants' use of the mobile application with the interface of the mobile epilepsy training program.
  During the monitoring phase, the Epilepsy Information Questions screen will be given once every 15 days, and the training module will be reopened automatically on missing or incorrect answers and the parent's information on this subject will be renewed.
  - At the end of the 3rd month, posttests (Parent Epilepsy Knowledge Scale for Parents and Parental Anxiety Scale for Seizures Scale) will be applied face-to-face.
  Interventions: Other: implementation of mobile epilepsy training program
- In the control group (No Intervention): - The purpose of the project will be shared with the parents in the control group, and the pre-tests Parent Epilepsy Knowledge Scale for Parents and Parental Anxiety Scale for Seizures Scale). will be applied.
  There is no structured training program in the outpatient functioning. Routine practice of the hospital; is the education and information provided by the physician to the family during the outpatient clinic.
  * At the end of the 3rd month, the final tests (Parent Epilepsy Knowledge Scale for Parents and Parental Anxiety Scale for Seizures Scale). will be applied face to face.
  * After the work is completed, the mobile application will be installed on the phones of the control group, the application will be taught and applied.

INTERVENTIONS:
Other: implementation of mobile epilepsy training program — Mobile epilepsy training program will be applied to the application group for 3 months.
  The mobile epilepsy training program developed within the scope of the thesis will be introduced to the parents in the application group and the participants will be uploaded to their phones via computer, and the use of the program will be taught in practice. In addition, the participants in the application group will be informed that the mobile epilepsy training program is not open to everyone during the research process, only the application group can use it. After the work is completed, the mobile application control group will be installed on the phones of the parents via computer, their application will be taught and applied.
  Arms: In application group; Mobile Epilepsy Training Program Impleme

SUMMARY:
Introduction: support to family and child related to epilepsy, controls or when they come for urgent reasons. Solutions must be found to ensure its continuity.

this support. The widespread use of the Internet today, e-health and health education is increasing day by day. Objective: The investigators research is planned to develop a mobile Epilepsy Training Program.

Parents with children diagnosed with epilepsy and assessing its effectiveness. Material and Method: The research is a randomized controlled experimental study.

An application was made to the Eskişehir Osmangazi University Clinical Research Ethics Committee and the ethics committee permission was obtained with the decision of 13.02.2020 dated 80558721-050.99-E.20230 and 2019-66 decision. Only volunteer participants will be included in the research. Its population study 3-6 years old children diagnosed with epilepsy Eskişehir City Hospital Child Neurology Outpatient Clinic between 01 September 2020 and 31 September 2021.

The sample of the research will consist of parents who meet the inclusion criteria.

research between these dates. Parents meeting research sample selection criteria The application was randomized as a control group according to the Parent Epilepsy Information Scale.

Application group; will use the mobile application the investigators prepared for the parent. Control group will consist of parents who follow the hospital's treatment protocol. The investigators study Completed with a total of 60 parents, 30 of whom are determined by power analysis group. Statistical analysis will be done with SPSS package program. Keywords: Child, Epilepsy, Parent Education, Mobile Application, Child Nurse

DETAILED DESCRIPTION:
Chronic disease is defined as a condition that deviates from the normal, results from pathological changes and leaves permanent insufficiency, continues for a long time, and requires special training, long-term care and treatment for the patient's rehabilitation. Epilepsy, one of the chronic diseases, is one of the most common neurological disorders in childhood.

The main goal in the treatment of epilepsy; It is based on the principle of ensuring seizure without harming the child's growth and development potential. In other words, controlling the seizures is to correctly identify the cause of the seizure and to help the child live a normal life.

According to the National Institute for Health and Clinical Excellence, the role of the epilepsy specialist nurse in epilepsy management is not limited to seizure control, but requires multi-dimensional care planning. It is an important nursing role to regulate the lifestyle and increase the compliance with the treatment to increase the patients' non-seizure. At the same time, the key roles of the epilepsy nurse include continuing cooperation with other healthcare team members, collaborating with the public and epilepsy-related organizations, and providing necessary information and educational support to families and children.

However, the support given to the family and the child is limited to the times that may come only with controls or for urgent reasons. Detailed solutions will be found to ensure the continuity of this support. Today, with the widespread use of the internet, healthcare education is increasing day by day. Web-based training applications prepared by professional experts are for information such as guidance, information and encouragement for patients with limited time and their parents. Participants phone contains at least one smartphone in almost every home in the internet age. there may be mobile applications to install.

With the use of mobile applications in health care services, it is seen that the quality of life of the patients and their relatives and the quality of health care services increase, but also contributes economically to health institutions.

The aim of the research is to develop and evaluate the effectiveness of the mobile epilepsy education program for parents with children diagnosed with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Can use and use Android based smart phone,
* Literate,
* Volunteers to participate in the study,
* Does not have any other chronic disease other than epilepsy,
* Parents with a child aged 3-6 years who are diagnosed with epilepsy at least six months ago (Tutar Güven, 2018) will be included in the study.

Exclusion Criteria:

* without an Android-based smartphone,
* IOS phone,
* Not capable of using mobile applications,
* Mentally disabled child
* Hearing impaired and do not speak Turkish
* Parents who are not willing to participate in the study will not be included in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Change in the knowledge of the applicant group about epilepsy disease | 12 weeks
  Change in the knowledge of the application group about epilepsy disease assessed with the Parent Epilepsy Information Scale "Parent Epilepsy Information Scale" will be filled in before and after the study (after 3 months) with the researcher, in order to measure the level of knowledge of parents about epilepsy.
  The high total score indicates that families have a high level of knowledge. Parents in the application group are expected to have an increased knowledge of epilepsy.
Change in anxiety of the applicant group about epilepsy disease | 12 weeks
  Change in anxiety level about epilepsy disease assessed with the The Parental Anxiety Scale for Seizures "The Parental Anxiety Scale for Seizures" will be filled with the face-to-face interview technique before and after the study (after 3 months) to determine the anxiety of the families of children with seizures. It is interpreted as the parental anxiety decreases as the score obtained from the scale increases.
  Anxiety levels of parents in the application group are expected to decrease.

CONTACTS AND LOCATIONS:
Overall Officials: DILEK SAYIK, PHD STUDENT, Principal Investigator — ESKİŞEHİR OSMANGAZİ UNIVERSITY INSTITUTE OF HEALTH SCIENCES
Locations (1):
- Eskisehir City Hospital, Odunpazari, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
With the mobile application, patients diagnosed with epilepsy and their parents / caregivers will be able to easily learn the correct information about epilepsy disease at any time (7/24) in any environment with a structured training program. Thanks to the mobile application, it will be possible to facilitate the compliance of diagnosis, follow-up and treatment in epilepsy disease. It is thought that mobile application will take place in child intensive care, child neurology and child clinics especially in the smartphones of children / parents / caregivers with epilepsy.
Supporting Information: Study Protocol
Time Frame: It will be shared after the study is finished (About 2 years later)
Access Criteria: It will be shared with child / parent / caregivers with epilepsy and child intensive care, child neurology and healthcare professionals working in child clinics.

REFERENCES:
- [Background] Fazlıoğlu, K., Hocaoğlu, Ç., & Sönmez F. M. Çocukluk Çağı Epilepsisinin Aileye Etkisi. Psikiyatride Güncel Yaklaşımlar, 2010; 2(2):189-205.
- [Background] Çavuşoğlu, H. Çocuk sağlığı hemşireliği, 10. Baskı. Ankara: Sistem Ofset Basımevi. 2011; 330-348.
- [Background] Dennis TA, O'Toole L. Mental Health on the Go: Effects of a Gamified Attention Bias Modification Mobile Application in Trait Anxious Adults. Clin Psychol Sci. 2014 Sep 1;2(5):576-590. doi: 10.1177/2167702614522228. PMID 26029490
- [Background] Falco-Walter JJ, Scheffer IE, Fisher RS. The new definition and classification of seizures and epilepsy. Epilepsy Res. 2018 Jan;139:73-79. doi: 10.1016/j.eplepsyres.2017.11.015. Epub 2017 Nov 28. PMID 29197668
- [Background] O'Conner-Von S. Coping with cancer: a Web-based educational program for early and middle adolescents. J Pediatr Oncol Nurs. 2009 Jul-Aug;26(4):230-41. doi: 10.1177/1043454209334417. Epub 2009 May 15. PMID 19448133
- [Background] Mo PK, Coulson NS. Developing a model for online support group use, empowering processes and psychosocial outcomes for individuals living with HIV/AIDS. Psychol Health. 2012;27(4):445-59. doi: 10.1080/08870446.2011.592981. Epub 2011 Aug 19. PMID 21854088
- [Background] National Institue for Health and Clinical Excellence. (2004). The diagnosis and management of the epilepsis in adults and children in primary and secondary care, NICE. Available from: http://www.nice.org.uk/nicemedia/pdf/CG020NICEguideline.pdf Access Date: 01.07.2019.
- [Background] Rodenburg R, Marie Meijer A, Dekovic M, Aldenkamp AP. Family predictors of psychopathology in children with epilepsy. Epilepsia. 2006 Mar;47(3):601-14. doi: 10.1111/j.1528-1167.2006.00475.x. PMID 16529629
- [Background] Scheffer IE, Berkovic S, Capovilla G, Connolly MB, French J, Guilhoto L, Hirsch E, Jain S, Mathern GW, Moshe SL, Nordli DR, Perucca E, Tomson T, Wiebe S, Zhang YH, Zuberi SM. ILAE classification of the epilepsies: Position paper of the ILAE Commission for Classification and Terminology. Epilepsia. 2017 Apr;58(4):512-521. doi: 10.1111/epi.13709. Epub 2017 Mar 8. PMID 28276062
- [Background] Zararsız, M. (2009). Epilepside güvenliğin sağlanmasına ilişkin çocuğa ve ebeveynlere verilen eğitimin etkinliğinin değerlendirilmesi, Yüksek Lisans Tezi, Mersin Üniversitesi Sağlık Bilimleri Enstitüsü, Mersin
- [Background] Wohlrab GC, Rinnert S, Bettendorf U, Fischbach H, Heinen G, Klein P, Kluger G, Jacob K, Rahn D, Winter R, Pfafflin M; Famoses Project Group. famoses: a modular educational program for children with epilepsy and their parents. Epilepsy Behav. 2007 Feb;10(1):44-8. doi: 10.1016/j.yebeh.2006.10.005. Epub 2006 Nov 27. PMID 17126082
- [Background] Tutar Güven, Ş. Ergen ve ebeveynlerine yönelik geliştirilen web tabanlı epilepsi eğitim programının etkinliğinin değerlendirilmesi, Doktora Tezi, Akdeniz Üniversitesi Sağlık Bilimleri Enstitüsü, Antalya. 2018